CLINICAL TRIAL: NCT01672996
Title: A Phase 1/2, Open Label, Randomized Study of Low Concentration Ioforminol Injections for Use in Contrast-Enhanced Abdominal Computed Tomography in Healthy Volunteers
Brief Title: Open Label, Randomized Study of Low Concentration Ioforminol Injections for Use in Abdominal CECT in Healthy Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Collaborators: Physician Reference Laboratory (Unknown); Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GE-145-004
Record Dates: First submitted 2012-08-09; First posted 2012-08-27 (Estimated); Results first posted 2014-03-03 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-04

CONDITIONS: Healthy
Keywords: Use in Abdominal; Contrast Enhanced; Computed Tomography; Optimize concentration; dosage of Ioforminol Injection
MeSH Terms: interventions — Iopamidol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 - Ioforminol 160mgI/mL (Experimental): Single administration of Ioforminol 160mgI/mL given to the subject.
  Interventions: Drug: Ioforminol 160 mgI/mL
- Arm 2 - Ioforminol 200mgI/mL (Experimental): Given as a single administration to the subject
  Interventions: Drug: Ioforminol 200 mgI/mL
- Arm 3 - Iopamidol 300mgI/mL (Active Comparator): Given as a single administration to the subject
  Interventions: Drug: Iopamidol 300 mgI/mL

INTERVENTIONS:
Drug: Ioforminol 160 mgI/mL — Given as s single administration to the subject
  Other Names: Ioforminol
  Arms: Arm 1 - Ioforminol 160mgI/mL
Drug: Ioforminol 200 mgI/mL — Given as a single administration to the subject
  Other Names: Ioforminol
  Arms: Arm 2 - Ioforminol 200mgI/mL
Drug: Iopamidol 300 mgI/mL — Given as a single administration to the subject
  Other Names: Iopamidol; Isovue 300; Isovue
  Arms: Arm 3 - Iopamidol 300mgI/mL

SUMMARY:
To optimize both the Ioforminol concentration and dosage(s) for CECT of the abdomen. To evaluate the safety and tolerability of low concentration Ioforminol Injections. Study recruits healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females between 18 and 50 years of age.
* The subject has a maximum abdominal circumference of 120 cm or less.

Exclusion Criteria:

* The subject has known Grade 3 or 4 allergic reaction/hypersensitivity to either iodine or any iodinated-based contrast agent or with history of multiple allergies (i.e., foods, pets, medications, etc).
* The subject has chronic renal insufficiency (estimated glomerular filtration rate [eGFR] <60 mg/dL) as measured at the screening visit.
* The subject is pregnant or breast-feeding.
* The subject has suspicion or diagnosis of hyperthyroidism or autonomously functioning thyroid nodule confirmed by T3, T4, and/or thyroid-stimulating hormone.
* The subject has severe liver or hematologic diseases (sickle cell disease or multiple myeloma), or immunodeficiency.
* The subject is taking metformin (e.g., Glucophage®) therapy.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2012-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rubin Sheng, MD, Study Director — GE Healthcare
Locations (1):
- GE Healthcare, Princeton, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1 - Ioforminol 160mgI/mL | Arm 2 - Ioforminol 200mgI/mL | Arm 3 - Iopamidol 300mgI/mL
Started | 30 | 30 | 6
Completed | 30 | 30 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1 - Ioforminol 160mgI/mL-1.0mL/kg: Ioforminol 160 mgI/mL: Given as s single administration to the subject.
  Dosing the Subject at 1.0mL/kg.
- Arm 1 - Ioforminol 160mgI/mL-1.5mL/Kg: Ioforminol 160 mgI/mL: Given as s single administration to the subject.
  Dosing the Subject at 1.5mL/kg.
- Arm 1 - Ioforminol 160mgI/mL-2.0mL/Kg: Ioforminol 160 mgI/mL: Given as s single administration to the subject.
  Dosing the Subject at 2.0mL/kg.
- Arm 2 - Ioforminol 200mgI/mL-1.0mL/kg: Ioforminol 200 mgI/mL: Given as a single administration to the subject.
  Dosing the Subject at 1.0mL/Kg
- Arm 2 - Ioforminol 200mgI/mL-1.5mL/kg: Ioforminol 200 mgI/mL: Given as a single administration to the subject.
  Dosing the Subject at 1.5mL/Kg
- Arm 2 - Ioforminol 200mgI/mL-2.0mL/Kg: Ioforminol 200 mgI/mL: Given as a single administration to the subject.
  Dosing the Subject at 2.0mL/Kg
- Arm 3 - Iopamidol 300mgI/mL-1.0mL/Kg: Iopamidol 300 mgI/mL: Given as a single administration to the subject.
  Dosing the Subject at 1.0mL/Kg
- Total: Total of all reporting groups
Arm/Group | Arm 1 - Ioforminol 160mgI/mL-1.0mL/kg | Arm 1 - Ioforminol 160mgI/mL-1.5mL/Kg | Arm 1 - Ioforminol 160mgI/mL-2.0mL/Kg | Arm 2 - Ioforminol 200mgI/mL-1.0mL/kg | Arm 2 - Ioforminol 200mgI/mL-1.5mL/kg | Arm 2 - Ioforminol 200mgI/mL-2.0mL/Kg | Arm 3 - Iopamidol 300mgI/mL-1.0mL/Kg | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 6 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 10 | 10 | 10 | 6 | 66
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 4 | 7 | 8 | 5 | 2 | 35
  Male | 5 | 6 | 6 | 3 | 2 | 5 | 4 | 31
Region of Enrollment [Number; unit: Participants]
  United States | 10 | 10 | 10 | 10 | 10 | 10 | 6 | 66

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Densities at Selected Regions in Contrast-enhanced CT Examination by Location (Abdominal Aorta), kVp 80 and Contrast Type (Ioforminol vs Iopamidol), Concentration (Ioforminol 160 or 200) and Dose Levels (1.0, 1.5, and 2.0mL/kg).
Description: Quantitative measurement of the radiographic density (as measured by Hounsfield Units (HU) ) at the abdominal aorta at the level of the celiac artery. The greater the contrast attenuation, the higher the HU.
Time Frame: Within 5 minutes after administration for either Ioforminol or Iopamidol.
Population: Evaluted 33 subjects using 80 kilovolt peak (kVp), a measure of the maximum electrical potential in kilovolts across an x-ray.
Measure: Mean (Standard Deviation); unit: Hounsfield Units
Arm/Group | Arm 1 - Ioforminol 160mgI/mL-1.0mL/kg | Arm 1 - Ioforminol 160mgI/mL-1.5mL/Kg | Arm 1 - Ioforminol 160mgI/mL-2.0mL/Kg | Arm 2 - Ioforminol 200mgI/mL-1.0mL/kg | Arm 2 - Ioforminol 200mgI/mL-1.5mL/kg | Arm 2 - Ioforminol 200mgI/mL-2.0mL/Kg | Arm 3 - Iopamidol 300mgI/mL-1.0mL/Kg
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 3
Hounsfield Units | 168 (41.0) | 261 (56.5) | 345 (30.7) | 341 (33.6) | 357 (30.1) | 365 (67.7) | 331 (53.7)

2. Secondary Outcome: Evaluate the Overall Safety of Ioforminol and Iopamidol Injections by Recording Treatment Emergent Adverse Events (TEAE).
Description: Recording the occurrence of treatment emergent adverse events (TEAE).
Time Frame: Up to 72 hours for safety monitoring post Ioforminol and Iopamidol administration.
Population: These are the numbers of Treatment Emergent Adverse Events (TEAE) and TEAEs related to Investigational Medicinal Product (IMP).
Measure: Number; unit: Adverse Events
Arm/Group | Arm 1 - Ioforminol 160mgI/mL-1.0mL/kg | Arm 1 - Ioforminol 160mgI/mL-1.5mL/Kg | Arm 1 - Ioforminol 160mgI/mL-2.0mL/Kg | Arm 2 - Ioforminol 200mgI/mL-1.0mL/kg | Arm 2 - Ioforminol 200mgI/mL-1.5mL/kg | Arm 2 - Ioforminol 200mgI/mL-2.0mL/Kg | Arm 3 - Iopamidol 300mgI/mL-1.0mL/Kg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 6
Adverse Events
  Any Treatment Emergent Adverse Events (TEAE) | 3 | 5 | 13 | 8 | 5 | 7 | 5
  Any Treatment Emergent Adverse Events-IMP | 2 | 5 | 13 | 8 | 5 | 7 | 5
  Intensity-Mild | 3 | 5 | 13 | 8 | 5 | 7 | 5
  Serious TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Withdrawals due to Adverse Events | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Deaths | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Radiographic Densities at Selected Regions in Contrast-enhanced CT Examination by Location (Abdominal Aorta), kVp 100 and Contrast Type (Ioforminol vs Iopamidol), Concentration (Ioforminol 160 or 200) and Dose Levels (1.0, 1.5, and 2.0mL/kg).
Description: as for outcome 1
Time Frame: Within 5 minutes after administration for either Ioforminol or Iopamidol.
Population: Evaluted 33 subjects using 100 kilovolt peak (kVp), a measure of the maximum electrical potential in kilovolts across an x-ray. tube.
Measure: Mean (Standard Deviation); unit: Hounsfield Units
Arm/Group | Arm 1 - Ioforminol 160mgI/mL-1.0mL/kg | Arm 1 - Ioforminol 160mgI/mL-1.5mL/Kg | Arm 1 - Ioforminol 160mgI/mL-2.0mL/Kg | Arm 2 - Ioforminol 200mgI/mL-1.0mL/kg | Arm 2 - Ioforminol 200mgI/mL-1.5mL/kg | Arm 2 - Ioforminol 200mgI/mL-2.0mL/Kg | Arm 3 - Iopamidol 300mgI/mL-1.0mL/Kg
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 3
Hounsfield Units | 191 (34.6) | 230 (40.2) | 212 (22.2) | 261 (37.7) | 246 (36.6) | 240 (49.4) | 257 (9.5)

ADVERSE EVENTS:
Time Frame: Up to 72 hours post Ioforminal or Iopamidol administration.
Arm/Group | Arm 1 - Ioforminol 160mgI/mL-1.0mL/kg | Arm 1 - Ioforminol 160mgI/mL-1.5mL/Kg | Arm 1 - Ioforminol 160mgI/mL-2.0mL/Kg | Arm 2 - Ioforminol 200mgI/mL-1.0mL/kg | Arm 2 - Ioforminol 200mgI/mL-1.5mL/kg | Arm 2 - Ioforminol 200mgI/mL-2.0mL/Kg | Arm 3 - Iopamidol 300mgI/mL-1.0mL/Kg
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/6
Other Adverse Events (participants affected / at risk) | 3/10 | 5/10 | 10/10 | 8/10 | 5/10 | 7/10 | 5/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 - Ioforminol 160mgI/mL-1.0mL/kg (N=10) | Arm 1 - Ioforminol 160mgI/mL-1.5mL/Kg (N=10) | Arm 1 - Ioforminol 160mgI/mL-2.0mL/Kg (N=10) | Arm 2 - Ioforminol 200mgI/mL-1.0mL/kg (N=10) | Arm 2 - Ioforminol 200mgI/mL-1.5mL/kg (N=10) | Arm 2 - Ioforminol 200mgI/mL-2.0mL/Kg (N=10) | Arm 3 - Iopamidol 300mgI/mL-1.0mL/Kg (N=6)
Nausea (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling Hot (General disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 5 (5)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 5 (5) | 9 (9) | 7 (7) | 5 (5) | 5 (5) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No